CLINICAL TRIAL: NCT06457100
Title: Comparison of the Effects of Perioperative Intravenous Infusions of Esmolol and Lidocaine on the Quality of Postoperative Recovery in Patients Undergoing Functional Endoscopic Sinus Surgery:A Randomized, Non-inferiority Trial
Brief Title: Esmolol Versus Lidocaine on the Quality of Postoperative Recovery in Patients Undergoing Functional Endoscopic Sinus Surgery
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Second People's Hospital of Huai'an (Other)
Responsible Party: Principal Investigator, Chenglan Xie, chief physician, The Second People's Hospital of Huai'an
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CXie
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Chronic Rhinosinusitis; Enhanced Recovery After Surgery
Keywords: Esmolol; Lidocaine; Postoperative recovery; Functional endoscopic sinus surgery
MeSH Terms: interventions — esmolol

STUDY DESIGN:
Intervention Model Description: In the esmolol group, 0.5 mg/kg esmolol was injected before the induction of anesthesia, and the injection was completed within 1 min, followed by continuous intravenous pumping of esmolol 50 ug/(kg-min) until the end of surgery.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The randomization sequence was generated by a computer and handed over in sealed opaque sequentially numbered envelopes. The envelope was opened by anaesthetist not involved in the study and drugs were dispensed as per the allocation card. The configured drugs were then handed over to experienced anaesthetists who were not aware of the subgroups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esmolol (Experimental): In the esmolol group, esmolol(2ml:0.2g) 0.5 mg/kg was given intravenously, pumped 1 min before induction of anesthesia, and then infused intravenously at 3.0 mg-kg-1 h-1 until the end of surgery.
  Interventions: Drug: Esmolol Injection
- Lidocaine (Active Comparator): In the lidocaine group, lidocaine(5ml:0.1g) 2.0 mg/kg was given intravenously, pumped 10 min before induction of anesthesia and then infused intravenously at 2.0 mg-kg-1 h-1 until the end of surgery.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Esmolol Injection — Before induction of anesthesia, 0.5 mg/kg of esmolol was pumped intravenously and infused within 1 minute, followed by a pumping rate of 3 mg/kg/h until the end of the procedure.
  Arms: Esmolol
Drug: Lidocaine IV — Before induction of anesthesia, 2 mg/kg of lidocaine was pumped intravenously and infused within 10 minute, followed by a pumping rate of 2 mg/kg/h until the end of the procedure.
  Arms: Lidocaine

SUMMARY:
Functional endoscopic sinus surgery (FESS) is one of the effective modalities for the treatment of chronic sinusitis, with the advantages of deep approach, light trauma, and less pain. However, because the operation area involves the nose, eyes and cranial region, the surrounding tissue structure is complex and rich in blood vessels and nerves, and the use of epinephrine, intraoperative tissue damage, nerve stimulation, and postoperative inflammation, edema, hemorrhage, and nasal cavity stuffing can cause patients' stress reaction and postoperative pain, resulting in patients' anxiety, depression, and sleep disorders, which can reduce the quality of early postoperative recovery, and affect the patients' rapid postoperative recovery. Esmolol is a selective β1-adrenergic receptor blocker with fast onset of action and short duration of action, which has the ability to reduce heart rate, blood pressure and myocardial protection. In recent years, several studies have found that esmolol not only reduces perianesthesia stress, but also reduces postoperative pain, decreases intraoperative and postoperative opioid requirements, and reduces the incidence of postoperative nausea and vomiting.In addition, intravenous lidocaine infusion has been shown to improve the quality of early postoperative recovery and accelerate postoperative recovery in patients with FESS.However, the dose of the drug administered is unclear and the range of safe infusion doses is narrow, requiring plasma concentration monitoring to prevent toxic reactions to local anesthetics. Its clinical application may lead to prolonged sinus bradycardia, increasing the cardiovascular risk of patients. Therefore, this study was designed to characterize the FESS procedure with the aim of determining that esmolol is not inferior to lidocaine in FESS in terms of the quality of postoperative recovery and is more advantageous in terms of controlling hemorrhage, guaranteeing a clear operative field, and the safety of the medication.

DETAILED DESCRIPTION:
In recent years, the concept of enhanced recovery after surgery (ERAS) has been widely used in the perioperative period of different diseases, but it has been rarely reported in patients undergoing functional endoscopic sinus surgery (FESS).

Therefore, the aim of this article was to compare the effects of esmolol and lidocaine on the quality of postoperative recovery in patients undergoing FESS. patients were randomly divided into: Group E: intravenous esmolol (0.5mg/kg for 1 min, followed by 3.0 mg/kg/h); Group L: intravenous lidocaine( 2.0 mg/kg for 10 min, followed by 2 mg/kg/h). The quality of recovery-15 (QoR-15) score was observed and compared between the two groups. Other parameters compared were: intraoperative field conditions, hemodynamic data, propofol, opioid and vasoactive drug dosage, Numeric rating pain scale (NRS), awakening and incidence of adverse effects.

The inclusion criteria were: age between 18 and 65 years, American Society of Anesthesiologists (ASA) classification I-II, FESS under general anesthesia. unsigned informed consent; major organ disease (such as cardiac, cerebral, pulmonary, hepatic, and renal disease); bradycardia and atrioventricular block; Bronchial asthma or history of bronchial asthma; patients with uncontrolled hypertension or hyperthyroidism; patients with diabetes mellitus or hearing impairment; those who were allergic to the drugs used in the experiment (such as esmolol or lidocaine) or experienced adverse drug reactions; pregnant and lactating women; those who had been taking long-term sedative or analgesic drugs, or who were chronically intoxicated; those with a history of psychiatric illnesses or those who had verbal communication disorders and were unable to comprehend the experimental content; and those who had a duration of surgery of more than 3 h; Patients who had a difficult airway during induction of anesthesia and required a change in routine intubation were excluded from this study.

Using a computer-generated randomization sequence and the sealed-envelope method, patients were randomly assigned to the esmolol and lidocaine groups in a 1:1 ratio. Patients, anesthesiologists, and investigators observing the results were unaware of the allocation of patient groups.

The patients were routinely fasted for 6 h and abstained from drinking for 2 h preoperatively. All patients were not anesthetized with premedication. After admission, patients were routinely administered oxygen by mask, peripheral venous access was opened and cardiac monitoring, including noninvasive blood pressure, pulse oximetry, electrocardiogram, body temperature and entropy index, was routinely performed. Both groups were routinely rapidly induced with midazolam 0.05 mg/kg, sufentanil 0.5 µg/kg, etomidate0.3 mg/kg, and rocuroniumbromide 0.6 mg/kg, respectively. Oxygen denitrification was administered for 3 min followed by endotracheal intubation and connection to a ventilator with pure oxygen of 1.0 L/min for respiratory control. Setting parameters: tidal volume 8～10 ml/kg, inspiratory ratio 1:2, control PETCO2 at 35～40 mmHg. Group E patients were pumped with saline for 10 min, followed by esmolol (0.5 mg/kg) for 1 min before the induction of anesthesia, and then continuous esmolol 3.0 mg/kg/h until the end of the surgery; Group L patients were pumped with lidocaine (2.0 mg/kg) for 10 min, followed by saline for 1 min before the induction of anesthesia , and then continuous lidocaine 3.0 mg/kg/h until the end of the operation. (both drugs were diluted to 20 ml with 0.9% saline). The appropriate depth of anesthesia (entropy index RE/SE 40-60) was maintained by adjusting the infusion rate of propofol and remifentanil. MAP was controlled at 60-75 mmHg, and vasoactive drugs (ephedrine, phenylephrine, and nitroglycerin) could be administered to regulate the blood pressure at the appropriate depth of anesthesia. After the operation, the patient was immediately transferred to the PACU. when the patient regained consciousness and could breathe on his own, the tracheal tube was removed. In the PACU, 30 mg of ketorolac tromethamine was administered intravenously to relieve analgesia if the patient's NRS score was ≥5 or if the patient required analgesia.

All scales were assessed by an independent anesthesiologist who was also unaware of the group assignment. The primary endpoint was QoR and was assessed at POD1 using the QoR-15 scale, a global measure of postoperative recovery. The QoR-15 scale consists of five dimensions, physical comfort, physical independence, emotional state, psychosocial support, and pain, with 15 items and a total score of 150 points. The higher the score, the better the quality of recovery. Secondary endpoints included: QoR-15 scores at preoperative (Preop) and POD2; NRS scores at 2 h, 4 h, 8 h, 24 h and 48 h postoperatively; MAP and HR at the time of patient admission, before induction, before intubation, immediately after intubation, 5 min after intubation, at the beginning of surgery, 5 min after the beginning of surgery, at the end of surgery, at the time of extubation, immediately after extubation, 5 min after extubation, and 30 min after extubation; the SF conditions (SSFQ is evaluated by the surgeon); intraoperative dosage of propofol, remifentanil, and vasoactive medications; the time to awakening and time to extubation (time from discontinuation to awakening and extubation); and the incidence of postoperative nausea, vomiting, and sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists (ASA) classification I-II
* Functional endoscopic sinus surgery under general anesthesia

Exclusion Criteria:

* Major organ disease (such as cardiac, cerebral, pulmonary, hepatic, and renal disease)
* Bradycardia and atrioventricular block
* Bronchial asthma or history of bronchial asthma
* Patients with uncontrolled hypertension or hyperthyroidism
* Patients with diabetes mellitus or hearing impairment
* Patients who were allergic to the drugs used in the experiment (such as esmolol or lidocaine) or experienced adverse drug reactions
* Pregnant and lactating women
* Patients who had been taking long-term sedative or analgesic drugs, or who were chronically intoxicated
* Patients with a history of psychiatric illnesses or those who had verbal communication disorders and were unable to comprehend the experimental content
* Patients who had a duration of surgery of more than 3 hours
* Patients who had a difficult airway during induction of anesthesia and required a change in routine intubation were excluded from this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-22 (Estimated)

PRIMARY OUTCOMES:
The quality of recovery-15（QoR-15） | Preoperative day、Postoperative day 1 、Postoperative day 2
  The QoR-15 scale is divided into five dimensions: physical comfort (5 items), self-care (2 items), psychological support (2 items), emotional state (4 items), and pain (2 items), with each item rated on a scale of 0-10, and the total score ranging from 0-150, with the higher the score the better the quality of recovery, and a score of 118 and above indicating surgery.

SECONDARY OUTCOMES:
surgical field quality score（SSMQ） | Immediately after surgery
  Surgical field quality was scored using the SSFQ scale, which can also be referred to as the Fromme Rating Scale, which consists of a scale of 1 to 5, corresponding to a score of 5 to 1. The higher the rating, the lower the score, and the worse the quality of the operative field.
Numeric rating scale（NRS） | 2 hours postoperative、4 hours postoperative、8 hours postoperative、24 hours postoperative、48 hours postoperative
  NRS is a rating used to assess a patient's level of pain, which is assessed by the patient based on self-perception on a scale from 0 to 10. A score of 0 represents no pain and a score of 10 represents the most pain.
Intraoperative propofol and remifentanil dosage | intraoperative
  The dosage of propofol and remifentanil was adjusted according to the depth of anesthesia during the operation, and propofol was maintained at a rate of 5~8 mg/kg/h, while remifentanil was maintained at 0.5~1.5 ug/kg/min.
incidence of adverse effects | Postoperative day 1 、Postoperative day 2
  the incidence of postoperative nausea, vomiting, and sore throat.
Intraoperative phenylephrine, atropine, nitroglycerin, ephedrine dosage | intraoperative
  Vasoactive drugs may be administered at an appropriate depth of anesthesia. When the mean arterial blood pressure(MAP) was >75 mmHg, 20 ug of nitroglycerin was given; when the MAP was less than 60 mmHg, 40 ug of phenylephrine was given preferentially, and 3 mg of ephedrine was given after the ineffective treatment; when the heart rate was less than 45 beats/minute, 0.5 mg of atropine was given.
Heart rate（HR） | admission to operating room、before induction of anesthesia、before intubation、immediately after intubation、start of surgery、end of surgery、at extubation
  perioperative hemodynamic fluctuations
Mean arterial blood pressure(MAP) | admission to operating room、before induction of anesthesia、before intubation、immediately after intubation、start of surgery、end of surgery、at extubation
  perioperative hemodynamic fluctuations

CONTACTS AND LOCATIONS:
Overall Officials: Xie chenglan, PhD, Study Director — The Affiliated Huaian Hospital of Xuzhou Medical University, Huai'an Second Hospital
Locations (1):
- The Affiliated Huaian Hospital of Xuzhou Medical University, Huai'an Second Hospital, Huaian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elaziz R A E A, Shaban S, Elaziz S A. Effects of Lidocaine Infusion on Quality of Recovery and Agitation after Functional Endoscopic Sinus Surgery: Randomized Controlled Study [J]. Open Journal of Anesthesiology, 2020, 10(12): 435-48.
- [Background] Bahr MP, Williams BA. Esmolol, Antinociception, and Its Potential Opioid-Sparing Role in Routine Anesthesia Care. Reg Anesth Pain Med. 2018 Nov;43(8):815-818. doi: 10.1097/AAP.0000000000000873. PMID 30216240
- [Background] Gelineau AM, King MR, Ladha KS, Burns SM, Houle T, Anderson TA. Intraoperative Esmolol as an Adjunct for Perioperative Opioid and Postoperative Pain Reduction: A Systematic Review, Meta-analysis, and Meta-regression. Anesth Analg. 2018 Mar;126(3):1035-1049. doi: 10.1213/ANE.0000000000002469. PMID 29028742
- [Background] Nair A. Esmolol: an avoidable agent for intraoperative use as an antinociceptive. Reg Anesth Pain Med. 2019 Jun;44(6):683. doi: 10.1136/rapm-2019-100429. Epub 2019 Mar 2. No abstract available. PMID 30826743
- [Background] Foo I, Macfarlane AJR, Srivastava D, Bhaskar A, Barker H, Knaggs R, Eipe N, Smith AF. The use of intravenous lidocaine for postoperative pain and recovery: international consensus statement on efficacy and safety. Anaesthesia. 2021 Feb;76(2):238-250. doi: 10.1111/anae.15270. Epub 2020 Nov 3. PMID 33141959
- [Background] Beaussier M, Delbos A, Maurice-Szamburski A, Ecoffey C, Mercadal L. Perioperative Use of Intravenous Lidocaine. Drugs. 2018 Aug;78(12):1229-1246. doi: 10.1007/s40265-018-0955-x. PMID 30117019
- [Background] Bajracharya JL, Subedi A, Pokharel K, Bhattarai B. The effect of intraoperative lidocaine versus esmolol infusion on postoperative analgesia in laparoscopic cholecystectomy: a randomized clinical trial. BMC Anesthesiol. 2019 Nov 4;19(1):198. doi: 10.1186/s12871-019-0874-8. PMID 31684867
- [Background] Moffatt DC, McQuitty RA, Wright AE, Kamucheka TS, Haider AL, Chaaban MR. Evaluating the Role of Anesthesia on Intraoperative Blood Loss and Visibility during Endoscopic Sinus Surgery: A Meta-analysis. Am J Rhinol Allergy. 2021 Sep;35(5):674-684. doi: 10.1177/1945892421989155. Epub 2021 Jan 21. PMID 33478255